CLINICAL TRIAL: NCT02952755
Title: A Randomized, Open-label, Crossover Study to Explore Drug-drug Interactions Between DWC20155 / DWC20156 and DWC20162 in Healthy Volunteers
Brief Title: Drug-Drug Interaction Study Between DWC20155 / DWC20156 and DWC20162 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWJ1366004
Record Dates: First submitted 2016-10-31; First posted 2016-11-02 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Healthy

ARMS (2):
- Study effect of DWC20162 on DWC20155/DWC20156 PK (Experimental): To study effect of DWC20162 on DWC20155/DWC20156 PK
  Interventions: Drug: Co-administration of DWC20155/DWC20156; Drug: DWC20162
- Study effect of DWC20155/DWC20156 on DWC20162 PK (Experimental): To study effect of DWC20155/DWC20156 on DWC20162 PK
  Interventions: Drug: Co-administration of DWC20155/DWC20156; Drug: DWC20162

INTERVENTIONS:
Drug: Co-administration of DWC20155/DWC20156
Drug: DWC20162

SUMMARY:
A randomized, open label, crossover study to explore drug-drug interactions between DWC20155 / DWC20156 and DWC20162 in Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria:

* Accepts healthy volunteers

Exclusion Criteria:

* Who has allergy to investigational product

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2016-12-12 (Actual); Study Completion 2016-12-20 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | 0 ~ 24 hours
Area under the time versus plasma concentration curve (AUC) | 0 ~ 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Bundang CHA Medical Center, Gyunggi, South Korea